CLINICAL TRIAL: NCT03086577
Title: Pain in Patients With Chronic Leg and Foot Ulcers - a Cross Sectional Study
Brief Title: Pain in Chronic Leg- and Foot Ulcers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College of Southeast Norway (Other)
Collaborators: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/1236 (REK)
Record Dates: First submitted 2017-02-15; First posted 2017-03-22 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Leg Ulcer; Pain
MeSH Terms: conditions — Leg Ulcer; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Leg ulcers are a significant cause of impaired functional ability and quality of life for approximately 1-2 percent of the population in western countries. Although pain seems to be one of the most devastating aspects of living with a chronic ulcer, research is limited and there is a lack of knowledge about wound-related pain characteristics. Little is known about prevalence, pain intensity, qualities, location, temporal fluctuations, to witch degree pain impact on physical- and psychosocial functioning, as well as relieving and exacerbating factors.

The overall purpose of this study is to investigate the prevalence and characteristics of wound related pain in patients with chronic leg ulcers. More specific research questions are: 1) What is the prevalence and characteristics of wound related pain in patients suffering from various types of persistent ulcers, 2) How do patients with different ulcer diagnoses report the quality of the wound related pain, 3) Is there any differences in wound pain characteristics among patients with different etiology leg ulcers, 4) How is the pain temporal pattern in patients with chronic leg- and foot ulcers, 5) What is the reported quality of life in patients with different ulcer diagnosis, and 6) Is there any association among pain characteristics, sleep and quality of life in patients with chronic leg/foot ulcers? The study has a non-experimental, explorative and descriptive approach. A cross-sectional questionnaire design will be used to explore patient's experience of wound-related pain.

The patients will be recruited at the outpatient clinic appointment and home-care nursing in Norway. Participants will fill out self-report questionnaires. The battery of questionnaires will obtain information about demographic data, pain characteristics, quality of life and sleep. Pain characteristics, quality of life and sleep will be assessed by using different questionnaires that has demonstrated high validity and reliability. In addition, the temporal pattern of pain will be assessed by asking the participants to fill out a form stating subjective level of pain (NRS) every hour during a typical day, and to mark times that they rest and sleep. Relevant information about the diagnosis/classification of ulcer, comorbidities, the ulcer management and pain management will be collected in a clinical examination.

DETAILED DESCRIPTION:
Design: The study has a non-experimental, explorative and descriptive approach. A cross-sectional questionnaire design, that provides quantitative data, will be used to explore patient's experience of wound-related pain.

Recruitment: Patients will be recruited from outpatient clinics and home-care nursing in Norway. Written informed consent will be obtained from all eligible patients who agree to participate.

The patients will be recruited at the outpatient clinic appointment. Those willing to participate will complete the questionnaire independently and return the questionnaire by mail in a pre-paid envelope. Furthermore, relevant information about the diagnosis/classification of ulcer, comorbidities, the ulcer management and pain management will be collected in a clinical examination, and by talking to the participants. The clinical examination will take place in relation to already scheduled dressing-change, in order to minimize the burden of participating in the study.

Based on clinical experience, and expert opinion, the research group have reason to believe that the ulcers can be classified in three main categories; ulcers with venous insufficiency as main perpetuating factor, ulcers with arterial insufficiency as main perpetuating factor, and ulcers with diabetes as the main perpetuating factor.

This study will not look at the effect-size of an intervention, or test a hypothesis. Therefore, the sample size is calculated based on the need to carry out the planed regression analysis to look at predictors of quality of life for patient with different etiology leg ulcers. In this study, quality of life will be a dependent variable, whereas pain, sleep, age, gender, wound area and possibly social status will be independent variables.

The sample size estimation is based on recommendations from statisticians and literature. The "rule of thumb" recommended indicates a study size of N> 104 + number of independent variables (here 6). This gives N> 110 in each group. The research group have chosen to set the sample size of 120 respondents in each group to take into account any dropouts. Three groups with 120 respondents result in a total sample size of 360 respondents.

The questionnaires Participants will fill out self-report questionnaires. The battery of questionnaires will obtain information about demographic and clinical data, pain characteristics, quality of life and sleep.

Demographic data: Information on age, gender, work situation, education, and living arrangements will be collected. This information will be used to describe the patient sample of the present study.

Clinical data: A research nurse will collect information about the patients' anamnesis and ulcer. Relevant information will be collected on the diagnosis/classification of ulcer, the ulcer management, and pain management. The measures included in this study are standardized measures in the clinic.

Diagnosis and classification of ulcer

The following data will be collected in order for the research-group to classify the different ulcers:

* The patients ulcer diagnosis (as stated by a medical doctor), the presumed causal factor (such as trauma or pressure), comorbidities, localization of the ulcer (on a body map), measure of wound size by multiplying the wounds width (millimeters at the widest) and height (millimeters at the highest).
* Clinical signs of wound-infection (critical colonization): Unusual/bad smell, visible pus, increased moisture, increased or changes in ulcer related pain, redness, swelling, heat, reduced general condition, and fever.
* Circulation of the leg will be assessed by palpation of ankle pulse. If no palpable pulse is found, the pulse will be assessed with Doppler. If unable to detect the pulse with Doppler, the Ankle-brachial pressure index will be calculated.
* Reduced sensibility will be assessed with the monofilament and tuning-fork tests for tactile and vibration sense.
* The presence of visible varices will be registered.
* A photograph of the ulcer and the lower leg and foot will be taken and used to classify the ulcers.
* Bothersome itch is assessed by asking the respondents.

Ulcer management: The research nurse will collect data on the ulcer management, such as the frequency of wound dressing change, if wet or dry dressing/treatment is used, and whether or not the patient has undergone ulcer debridement or revision surgery during the last week. Furthermore, if the patient is recruited at an outpatient clinic, the patient is asked whether this is the first consultation at the clinic.

Pain management: Both medical and non-medical treatment for pain is registered. It will be differentiated whether the pain management is aimed at ulcer pain or other types of pain that the patients may suffer from.

Characteristics of wound-related pain Pain intensity: The 0 - 10 Numeric Rating Scale (NRS) for pain is a one-dimensional measure of pain intensity.

Pain qualities: The Short Form McGill Pain Questionnaire (SF-MPQ) will be used to assess different qualities of the subjective pain experience. The aim of this questionnaire is to capture pain as a multidimensional phenomenon, recognizing the shortcomings of simple pain intensity scales.

The Brief Pain Inventory (BPI): BPI provides information about the location, intensity, treatment and impact of pain.

Temporal pattern of pain: There are no questionnaire available adapted for assessment of pain pattern for use in self-report at one set time. The research group has designed and will test a one-dimensional tool to assess the pattern of wound pain. The first part of the tool is based on the last item of the Pain Quality Assessment Scale where the respondents select one of tree statements reflecting intermittent pain, variable pain and stabile pain. The second part of the tool includes a graph where the respondents indicate subjective level of pain (0 - 10 NRS) every hour during a typical day. Pertaining to level of pain, the participants also mark specific times during the day spent in activity, resting, and sleeping.

Localization of wound-related pain: The respondents will be asked about the location of wound-related pain, and can choose among multiple alternative options, such as directly in the wound or wound-bed, in the wound-edges, in the skin surrounding the wound, in the entire foot, and in the entire leg. The respondents can also write in own words where the wound pain is located.

Quality of life Will be assessed using The EuroQol-5D (EQ-5D) which is a standardized instrument developed by the EuroQol Research Foundation for use as a measure of health outcome applicable to a wide range of health conditions.

Sleep The Insomnia Severity Index (ISI) is a brief self-report instrument measuring the patient's perception of sleep. The ISI targets the subjective symptoms and consequences of insomnia as well as the degree of concerns or distress caused by those difficulties.

Analyses The data will be analyzed with appropriate parametric and nonparametric tests using Statistical Package for the Social Sciences for Windows. The data will be analyzed using means, standard deviations, correlation coefficients, analysis of variance (ANOVA) and regression analyses.

The photographs and clinical ulcer data will be evaluated by the research-group in order to categorize the ulcers, based on predefined criteria for three etiology groups.

Ethical considerations This study is approved by the Regional Committees for Medical and Health Research Ethics in Norway (region south-east). This should assure that the study follows all necessary ethical considerations regarding cross-sectional quantitative research design. Furthermore, the study is reported to the Data Inspectorate. Application for permission to recruit participants has also been sent to the Head of the department in the different clinics and community nursing services where patients will be recruited.

Participation in the study will be voluntary, and there will be no obligation to participate or "penalty" or consequences for not participating. Patients will receive written and oral information about study participation. An introductory letter that describes the purpose and nature of the study and confidentiality of the data, as well as a written consent, form will be handed out to potential participants. Patients willing to participate need to sign the consent form before receiving the questionnaire. Confidentiality will be maintained through coding of participants and removal of identifiers at an early stage in data analysis. Completed questionnaires and codebooks will be stored separately and according to rules and regulations set by the Ethics Committee and the involved hospital and community nursing services. The completed questionnaires will be stored in locked and fire-safe safes. Digital copies of data will be saved on research-servers at the University College of Southeast-Norway (HSN).

The photographs taken of the patients' ulcers will not contain information that can identify the patients. The study nurse will take the photo so that it only visualizes the wound and lower leg/foot. The photo will be allocated the patients study-identification number, and saved electronically on the research server at the HSN. No hard-copies of the photo will be stored.

ELIGIBILITY:
Inclusion Criteria:

* Leg- or foot ulcer that has persisted for more than 6 weeks

Exclusion Criteria:

* Psychological and cognitive restrictions that prohibit from providing informed consent, reading or writing disabilities
* Inability to participate due to physical/psychological challenges, and inability to differentiate wound-related pain from other types of pain in the lower extremities.
* The following ulcer-diagnosis will be excluded: Burn-ulcer, cancer-ulcer, radiation-ulcer, immunological ulcers and vasculitis ulcers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult persons, with a leg- or foot ulcer that has persisted for more than 6 weeks, and are treated in outpatient clinics and home-care nursing services in Norway.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-02-21 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity - Numeric Rating Scale (NRS) | Through study completion, an average of 3 years
  One-dimensional measure of pain intensity.

SECONDARY OUTCOMES:
Sleep assessment - The Insomnia Severity Index (ISI) | Through study completion, an average of 3 years
  ISI is a brief instrument measuring the patient's perception of their sleep
Quality of life - The EuroQol-5D (EQ-5D) | Through study completion, an average of 3 years
  Measure of health outcome (walking, personal hygiene, daily function, pain and discomfort, anxiety and depression)
Quality of pain - The Short Form McGill Pain Questionnaire (SF-MPQ) | Through study completion, an average of 3 years
  SF-MPQ will be used to assess different qualities of the subjective pain
Brief Pain Inventory (BPI) | Through study completion, an average of 3 years
  BPI provides information about the location, intensity, treatment and impact of pain.
Localization of pain, Body map for localization of pain | Through study completion, an average of 3 years
  The respondents will be asked to locate their pain my marking localization on a body map. In addition, the respondents will be asked about the location of their wound-related pain, and can choose among multiple alternative options, such as directly in the wound or wound-bed, in the wound-edges, in the skin surrounding the wound, in the entire foot, and in the entire leg. The respondents can also write in their own words where the wound pain is located.
Temporal pattern of pain | Through study completion, an average of 3 years
  Based on the last item of the Pain Quality Assessment Scale where the respondents select one of tree statements reflecting intermittent pain, variable pain and stabile pain.
Variation of pain intensity throughout the day | Through study completion, an average of 3 years
  A graph where the respondents indicate their level of pain (0 - 10 NRS) every hour during a typical day

CONTACTS AND LOCATIONS:
Overall Officials: Tone M Ljosaa, Phd, Principal Investigator — Univerity Collage of Southeast Norway
Locations (1):
- Vestre Viken, Drammen, Buskerud, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Oversight authorities presentation of the study — https://helseforskning.etikkom.no/prosjekterirek/prosjektregister/prosjekt?p_document_id=710803&p_parent_id=745298&_ikbLanguageCode=n